CLINICAL TRIAL: NCT03931876
Title: A Placebo Controlled, Double Blind, Single Ascending Dose Study of AV-006 in Healthy Subjects
Brief Title: A Single Ascending Dose Study of AV-006 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arixa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Arixa-AV-006-01
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebos
- Active (Active Comparator): AV-006
  Interventions: Drug: AV-006

INTERVENTIONS:
Drug: Placebos — Single ascending dose administration
  Arms: Placebo
Drug: AV-006 — Single ascending dose administration
  Arms: Active

SUMMARY:
Characterization of the single dose pharmacokinetics of AV-006 in healthy male and female subjects. Description of safety and tolerability of AV-006 in healthy subjects

DETAILED DESCRIPTION:
The present study is a first in human study of an avibactam prodrug to be administered orally. Avibactam is the β-lactamase inhibitor (BLI) component of the intravenous antibiotic AVYCAZQR (ceftazidime avibactam), approved in the US in 2015 to treat resistant Gram-negative infections. Avibactam is a non-β-lactam BLI without intrinsic antibacterial activity. Avibactam binds covalently with bacterial β-lactamases thereby preventing hydrolysis and inactivation of the partner β-lactam antibiotic.

Arixa and others have shown that that avibactam (the product of AV-006) restores the susceptibility of many oral β-lactam antibiotics against broad panels of clinical Enterobacteriaceae isolates that produce β-lactamases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 18-55 (inclusive).
2. Good general health, with no significant medical history. Subjects must have no clinically significant abnormalities on physical examination at screening, and/or before administration of study drug
3. Body weight ≥ 50 kg at the screening visit
4. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
5. Has laboratory values (clinical chemistry and hematology) within the normal reference range. Deviations from this range may be acceptable if they are considered not clinically significant' (NCS) by the PI
6. Women of childbearing potential may be enrolled if one of the following criteria applies:

   1. Must be using two methods of contraception, consisting of (1) a highly-effective method associated with a < 1% failure rate when used correctly and consistently (e.g. hormonal contraception methods associated with suppression of ovulation or an IUD) and (2) partner use of a condom. Contraception should have been used for at least one month prior to study entry, the subject must have maintained a normal menstrual pattern for the three months prior to study entry and have a negative pregnancy test (urine) at the time of admission to the unit. Women must be willing to continue this contraception for 45 days following administration of study drug
   2. Is abstinent from heterosexual intercourse where this is consistent with the participant's usual and preferred lifestyle
   3. Is monogamous with a vasectomized partner (>3 months prior)
   4. Is postmenopausal (i.e., no cycle for at least the previous 12 months, is of menopausal age (> 45 years) and has a negative pregnancy test (urine) both at Screening and Day -1)
   5. Is surgically sterilized (confirmed by medical record review)
   6. Has had a total hysterectomy a minimum of 3 months prior to dosing on Day 1 (confirmed by medical record review)
7. Males who are sexually abstinent may be enrolled or, if sexually active, may be enrolled if one of the following criteria applies:

   1. Has had a vasectomy (>3 months prior to study entry, confirmed by medical record review)
   2. Using condoms and whose partner is using an acceptable form of contraception (IUD, oral contraceptives, birth control patch or vaginal ring, injectable or implanted contraceptives, or tubal ligation [surgical sterilization]) from Day -1 to 90 days after study drug administration
8. Understands the study procedures and agrees to participate in the study by giving written informed consent
9. Is a non-smoker (i.e. fewer than 4 cigarettes in 12 weeks prior to screening) Able and willing to attend the necessary visits to the study center

Exclusion Criteria:

1. Blood donation or recipient of blood transfusion in previous 30 days.
2. History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
3. History of neoplastic disease (except adequately-treated non-melanomatous skin carcinoma)
4. Mentally or legally incapacitated, ie has significant emotional problems at the time of Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder within the last 5 years
5. Fever (body temperature >38◦C) or symptomatic viral/bacterial infection or use of antibiotics within 2 weeks prior to Screening
6. Resting blood pressure (BP) >140/90 mmHg or heart rate (HR) >100 beats per minute at Screening or at Day -1 (vital signs to be taken with subject in semi- recumbent position)
7. Clinically significant abnormality on ECG performed at the Screening Visit or prior to administration of the initial dose of study drug. (Screening and predose ECG conduction intervals (corrected for heart rate) must be within the normal range).
8. Clinically significant laboratory abnormalities. Impaired renal function (which should be determined on the Screening day only) to be estimated using creatinine clearance (CrCl) of <80 mL/minute based on the appropriate formula for calculation of CrCL [calculation to be performed by laboratory responsible]
9. Positive test for hepatitis C antibody, hepatitis B surface antigen, or human immunodeficiency virus (HIV) antibody at Screening
10. Participants with a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol, amphetamines, benzodiazepines, opiates and cocaine)
11. Participants with a history of substance abuse or dependency or history of recreational IV drug use (by self-declaration)
12. Alcohol consumption >14 alcohol units per week. (One unit of alcohol is 10 ml, in- formation on calculation the content of drinks is provided at: http://www.alcohol.gov.au/internet/alcohol/publishing.nsf/Content/standard)
13. Unable to refrain from or anticipates the use of any medications, including prescription and non-prescription drugs and herbal remedies (such as St. John's Wort [Hypericum perforatum]), beginning 14 days (or 5 half-lives, whichever is longer) before administration of the initial dose of study drug and continuing throughout the study until the final study visit. There may be certain medications that are permitted at the discretion of the Investigator and Sponsor (including paracetamol/acetaminophen, medications for the treatment of AEs following administration of study drug
14. Subjects who are unlikely to comply with the study protocol or, in the opinion of the investigator, would not be a suitable candidate for participation in the study.
15. Have participated in any other investigational drug trial within 30 days of dosing in the present stud
16. Known intolerance of or sensitivity to avibactam

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-24 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events, vital signs data, ECGs, clinical laboratory tests of AV-006 following oral administration | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, PhD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No